CLINICAL TRIAL: NCT05458440
Title: Human Leucocytes Bank From COVID-19 Cured Patients With a Cellular Immunity Against SARS-CoV-2 :Raw Material for the Preparation of an Anti-SARS-CoV-2 Cellular Immunotherapy
Brief Title: Bank of Human Leukocytes From COVID-19 Convalescent Donors With an Anti-SARS-CoV-2 Cellular Immunity
Acronym: COVIBank
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, LEFEVRE Benjamin, Doctor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A02179-32
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Cellular Immunotherapy; Viral specific T cells; Bank
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Covid-19 Convalescent donors (Other): The protocol will be explained during hospitalisation for each donor infected by SARS-CoV-2. If they agree, they will be included before they leave hospital. Few weeks later, if they have no exclusion criteria, they will consult in the hemapheresis department of the Nancy University hospital. After medical exams, a whole blood bag and blood samples will be taken with the aim to establish a bank of cryopreserved human leucocytes as a raw material for the generation of a T-Lymphocyte immunotherapy.
  Interventions: Other: Generation of a biobank allowing the cryopreservation of leucocytes from COVID19 convalescent donors

INTERVENTIONS:
Other: Generation of a biobank allowing the cryopreservation of leucocytes from COVID19 convalescent donors — The investigators aim to demonstrate that it is possible to implement a biobank of leucocytes from convalescent donors that could be used as raw material to generate anti-SARS COV-2 viral specific T cells. The protocol will be explained during hospitalisation for each donor. If they agree, they will be included before they leave hospital. Few weeks later, if they have no exclusion criteria, they will consult in the hemapheresis department of the Nancy University hospital. After medical exams, a whole blood bag and blood samples will be taken with the aim to establish a bank of cryopreserved human leucocytes as a raw material for the generation of a T-Lymphocyte immunotherapy.

SUMMARY:
The SARS-CoV-2 identified in China in January 2020 is the cause of an unprecedented pandemic. The SARS-CoV-2 and each viral variant are responsible of a respiratory infectious disease, which can be asymptomatic. Nevertheless, a part of infected patients will experiment serious forms associated with a high mortality rate. Most serious forms present with lymphopenia and a functional exhaustion of speicifci T lymphocytes. Several studies showed that these quantitative and qualitative lymphocyte abnormalities are associated with unfavourable patients' outcome. The investigators hypothesized that the use of anti-viral T lymphocytes from convalescent COVID 19 donors could be helpful to improve the prognosis of COVID-19 serious forms. This study aims to demonstrate the feasibility of setting up a biobank that could allow the preservation and production of a cellular immunotherapy specific to SARS-CoV-2.

DETAILED DESCRIPTION:
Patients who meet the donor selection criteria during their hospitalization for a COVID-19 infection in the Infectious and Tropical Diseases Department of the University Hospital of Nancy will be informed of the study.

Recovery generally occurs within 14 days of the date of infection (D0) corresponding to the date of appearance of the first symptoms of the infection. This is characterized by the disappearance of patent clinical symptoms such as fever and chills and, for patients hospitalized for O2 requisition, in the cessation of oxygen therapy.

A medical visit will be scheduled within 28 to 64 days after the beginning of the SARS-Cov-2 infection (D28 to D64) with the department of hemapheresis of the Nancy university hospital for the collection of a whole blood bag.

Forty-eight hours before this medical appointment (D26 to D62), the patients included in the study will be contacted again by phone to ensure that they do not present a contraindication (fever, appearance of new symptoms since healing and/or feverishness) to the continuation of the study.

In absence of contraindications, the medical appointment is maintained. During the medical appointment, the regulatory infectious markers for (i) HIV, (ii) HTLV, (iii) hepatitis, (iv) syphilis, (v) EBV, (vi) CMV and (vii ) toxoplasmosis will be sought.

The following will also be collected:

(i) a bag of whole blood (450 ml); (ii) 2 x 7 ml dry tubes for serological analyses; (iii) 3 x 7 ml EDTA tubes for DGV; (iv) 3 tubes of 5 ml on lithium heparin for the Elispot test and (v) 1 tube of EDTA of 7 ml for HLA typing. The blood bags will be transported to the Nancy University Hospital Cell Therapy unit (UTCT). The whole blood samples go into production and undergo a density gradient separation in order to isolate mononuclear cells before cryopreservation.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalised for proved SARS-CoV-2 infection in the infectious disease unit of the Nancy University Hospital who received a comprehensive information about the study, and accepted to participate
* Patient who has an active cellular immunity against SARS-CoV-2 (biological definition: Elispot IFNgamma : > 50 SFC/106 PBMC)

Exclusion Criteria:

* Patient hospitalised in Intensive car unit
* Patient with haemoglobin < 10 g/dl
* Patient who take hypertension medication
* Patient with cardiovascular history: Valvulopathy, conduction rythm disorders, arterial vascular insufficiency, congenital anomalies
* Patient with auto-immune disease
* Patient with medical history of solid or hematopoietic graft
* Patient with active malignant disease (haematological or neoplasm) or considered in remission since less than 2 years
* Patient with psychiatric disorders
* Patient subject to a legal protection measure.
* Patient with proved infectious disease
* Asplenic patient
* Pregnant or breastfeeding woman
* Woman without contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
To build a biobank of convalescent donors T-lymphocytes samples | 12 months
  The mononuclear cells of convalescent COVID-19 patients meeting the criteria will be cryopreserved in the bank (feasability study)

SECONDARY OUTCOMES:
To determine the HLA-type of each leucocyte samples in the bank by DNA-sequencing | 12 months
  The investigators will determine for each patient's biological sample the type of HLA (A, B, DRB1). For this step, a DNA sequencing with new generation sequencing (Illumina MiniSeq) will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU-Nancy - Hopitaux de Brabois - Batiment Philippe Canton, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No